CLINICAL TRIAL: NCT01925781
Title: e-Cigarettes Versus Nicotine Replacement Therapy for Smoking Cessation
Brief Title: e-Cigarettes Versus NRT Gum for Smoking Cessation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: IND required
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-16684
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Nicotine Addiction; Smoking Cessation
Keywords: Smoking Cessation; Nicotine Addiction; e-Cigarette; electronic nicotine delivery device; electronic cigarette; nicotine replacement therapy
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Vaping | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- e-Cigarette (Experimental): STAM 1100mAh CE4 eGo Clearomizer e-Cigarette
  Interventions: Other: STAM 1100mAh CE4 eGo Clearomizer
- Nicotine polacrilex (Active Comparator): Nicotine Replacement gum
  Interventions: Drug: Nicotine polacrilex

INTERVENTIONS:
Drug: Nicotine polacrilex — 2 mg and 4 mg gum will be used according to the FDA approved product labelling
  Other Names: Nicotine Gum
  Arms: Nicotine polacrilex
Other: STAM 1100mAh CE4 eGo Clearomizer
  Other Names: e-Cigarette; electronic nicotine delivery device
  Arms: e-Cigarette

SUMMARY:
This is a randomized trial comparing electronic cigarettes (e-Cigarettes) to nicotine gum for smoking cessation. Participants will be randomly assigned to either e-cigarette use or nicotine gum use during a quit attempt. All participants will have a one hour meeting with a tobacco treatment specialist to develop a quit plan and set a quit date. Quit status will be determined at 12 weeks after the quit date. Continued use of nicotine replacement (either e-Cigarette or nicotine gum) and satisfaction with the treatment assignment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Smokes at least five cigarettes per day
* No current or previous regular use of e-cigarettes
* Ready to quit smoking

Exclusion Criteria:

* Use of smokeless or pipe tobacco
* Smoke more than 40 cigarettes per day
* Pregnant or breastfeeding
* Unable to chew gum due to dental or jaw problems
* Myocardial infarction (heart attack) within the previous 12 months
* Hypersensitivity to propylene glycol or nicotine gum

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Arouni, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | e-Cigarette | Nicotine Polacrilex
Started | 5 | 5
Completed | 3 | 1
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | e-Cigarette | Nicotine Polacrilex | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 42 [26 to 62] | 44 [34 to 61] | 43 [26 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Sustained Abstinence
Description: No smoking at 12 weeks after the predetermined quit date with a 5 day grace period. Self-report will be biochemically confirmed with expired carbon monoxide (CO) and salivary cotinine.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | e-Cigarette | Nicotine Polacrilex
Number analyzed (Participants) | 3 | 1
participants | 0 | 1

2. Secondary Outcome: Point Prevalence Abstinence
Description: No smoking in the previous 7 days. Self report will be biochemically confirmed with expired CO and salivary cotinine.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | e-Cigarette | Nicotine Polacrilex
Number analyzed (Participants) | 3 | 1
participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | e-Cigarette | Nicotine Polacrilex
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | e-Cigarette (N=5) | Nicotine Polacrilex (N=5)
Throat dry/irritated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes